CLINICAL TRIAL: NCT02057757
Title: A Randomized Double-Blind Phase 2 Study Comparing the Efficacy, Safety, and Tolerability of Nitazoxanide Versus Placebo in Addition to Standard Care for the Treatment of Hospitalized Subjects With Severe Acute Respiratory Illness
Brief Title: Nitazoxanide Versus Placebo for the Treatment of Hospitalized Subjects With Severe Acute Respiratory Illness
Acronym: NTZ-SARI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Mexican Emerging Infectious Diseases Clinical Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTZ-SARI
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Severe Acute Respiratory Illness
MeSH Terms: interventions — nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitazoxanide (NTZ) (Experimental): Participants will receive NTZ for 5 days. Participants younger than 12 years will receive an oral suspension formulation of NTZ; participants 12 years and older will receive NTZ tablets.
  Interventions: Drug: Nitazoxanide
- Placebo (Placebo Comparator): Participants will receive placebo for 5 days. Participants younger than 12 years will receive an oral suspension formulation of placebo; participants 12 years and older will receive placebo tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitazoxanide — Participants 1 to 3 years old: 5 mL oral suspension (100 mg NTZ) every 12 hours for 5 days.
  Participants 4 to 11 years old: 10 mL oral suspension (200 mg NTZ) every 12 hours for 5 days.
  Participants 12 years and older: two 300-mg NTZ tablets orally twice daily for 5 days.
  Other Names: NTZ
  Arms: Nitazoxanide (NTZ)
Drug: Placebo — Participants 1 to 3 years old: 5 mL placebo oral suspension every 12 hours for 5 days.
  Participants 4 to 11 years old: 10 mL placebo oral suspension every 12 hours for 5 days.
  Participants 12 years and older: two placebo tablets orally twice daily for 5 days.
  Other Names: PCB
  Arms: Placebo

SUMMARY:
Respiratory viruses are a significant cause of hospitalization for respiratory tract infections. This study will evaluate the safety, effectiveness, and tolerability of nitazoxanide (NTZ) in treating severe acute respiratory illness (SARI) in people who are hospitalized.

DETAILED DESCRIPTION:
Respiratory viral infections are one of the most common causes of illness in the world. These infections are major causes of SARI and can lead to severe outcomes, including hospitalization and death. NTZ is a medication that is approved in the United States and Mexico to treat gastrointestinal parasitic diseases. This study will evaluate the use of NTZ to treat SARI. The purpose of this study is to evaluate the safety, effectiveness, and tolerability of NTZ, in combination with standard care, in treating SARI in people who are hospitalized.

Participants will be hospitalized and study entry assessments will include medical assessments, blood collection, and a nasopharyngeal swab or wash. Participants will then be randomly assigned to receive NTZ or placebo for 5 days. Participants younger than 12 years will receive an oral suspension formulation of NTZ or placebo; participants 12 years and older will receive NTZ or placebo tablets. All participants will also receive standard of care treatment for acute severe viral respiratory infections, which may include antibiotics and/or treatment for influenza. They will be discharged from the hospital based on their doctors' recommendations. Participants will record their temperature and symptoms in a daily diary, which will be reviewed by study staff during study visits. Follow-up visits will occur on Days 3, 7, 14, and 28, and may occur as inpatient or outpatient visits. These visits may include the same assessments that occurred at baseline, as well as physical examinations, depending on the visit. Participants who are still hospitalized at Day 28 will be followed by study staff until they are discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to performance or initiation of any study procedures
* Age greater than or equal to 12 months of age (no upper age limit)
* Influenza-like illness (ILI), defined as (all of the following):

  * Onset of fever greater than or equal to 38°C (or hypothermia less than 36°C)
  * New or worse cough or sore throat
  * New or worse shortness of breath or difficulty breathing
* Onset of illness no more than 5 days before screening defined as when the participant experienced at least 1 respiratory symptom, constitutional symptom, or fever
* Hospitalization for ILI (decision for hospitalization will be up to the individual treating clinician), with anticipated hospitalization for more than 24 hours
* One of the following to avoid pregnancy:

  * Females who are able to become pregnant (i.e., are not postmenopausal, have not undergone surgical sterilization, and are sexually active with men) must agree to use at least 1 effective form of contraception from the date of informed consent through Day 28 of study
  * Males who have not undergone surgical sterilization and are sexually active with women must agree to use condoms or have a partner use at least 1 effective form of contraception through Day 28 of study

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Clinical suspicion that etiology of illness is primarily bacterial in origin
* Prior treatment with antivirals (e.g., oseltamivir) for the current illness for more than 24 hours
* Unable to take oral medications (adults must tolerate tablets, children must tolerate suspension)
* Unable to tolerate oral food/fluids (absorption is significantly better with food)
* Prior treatment with any investigational drug therapy within 30 days prior to screening
* Known sensitivity to NTZ or any of the excipients comprising the NTZ tablets
* Prior NTZ use within 1 week
* Self-reported history of chronic kidney disease or impaired renal function (no blood or urine kidney function laboratory testing will be done prior to enrollment, but intent is to exclude disease severe enough to cause estimated creatinine clearance [CrCl] less than 30)
* Self-reported history of liver disease (no blood laboratory testing will be done prior to enrollment, but intent is to exclude disease severe enough to cause cirrhosis or total bilirubin greater than 2, aspartate aminotransferase [AST]/alanine aminotransferase [ALT] greater than 3 times the upper limit of normal [ULN])
* Presence of any pre-existing illness that, in the opinion of the investigator, would place the participant at an unreasonably increased risk through participation in this study
* Participants who, in the judgment of the investigator, will be unlikely to comply with the requirements of this protocol
* The onset of SARI occurs after hospitalization
* Hospitalized for any reason for greater than 48 hours prior to enrollment
* Participants previously enrolled in this study
* Prior hospital discharge within 30 days
* Known chronic respiratory infection (e.g., tuberculosis, atypical mycobacterial infections)

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2014-02; Primary Completion 2017-05 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Guerrero Almeida, M.D., Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Ana Gamiño, M.D., Study Chair — Hospital Infantil de Mexico Federico Gomez; Arturo Galindo Fraga, M.D., Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Sarbelio Moreno, M.D., Principal Investigator — Hospital Infantil de Mexico Federico Gomez; Javier Araujo Melendez, M.D., Principal Investigator — Hospital Central "Dr. Ignacio Morones Prieto"; Alejandra Ramirez Venegas, M.D., Principal Investigator — Instituto Nacional de Enfermedades Respiratorias; Beatriz Llamosas Gallardo, M.D., Principal Investigator — Instituto Nacional de Pediatria; Yuri Roldan Aragon, M.D., Principal Investigator — Hospital General Dr. Aurelio Valdivies
Locations (6):
- Mexico (6):
  - Instituto Nacional de Pediatria, Coyoacán
  - Hospital General Dr. Aurelio Valdivieso, Oaxaca City
  - Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City
  - Hospital Infantil de Mexico Federico Gomez, Tamaulipas
  - Instituto Nacional de Ciencias medicas y Nutricion Salvador Zubiran, Tlalpan
  - Instituto Nacional de Enfermedades Respiratorias, Tlalpan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gamino-Arroyo AE, Guerrero ML, McCarthy S, Ramirez-Venegas A, Llamosas-Gallardo B, Galindo-Fraga A, Moreno-Espinosa S, Roldan-Aragon Y, Araujo-Melendez J, Hunsberger S, Ibarra-Gonzalez V, Martinez-Lopez J, Garcia-Andrade LA, Kapushoc H, Holley HP, Smolskis MC, Ruiz-Palacios GM, Beigel JH; Mexico Emerging Infectious Diseases Clinical Research Network (LaRed). Efficacy and Safety of Nitazoxanide in Addition to Standard of Care for the Treatment of Severe Acute Respiratory Illness. Clin Infect Dis. 2019 Nov 13;69(11):1903-1911. doi: 10.1093/cid/ciz100. PMID 30753384

RESULTS

PARTICIPANT FLOW:
Groups:
- Nitazoxanide (NTZ): Participants will receive NTZ for 5 days. Participants younger than 12 years will receive an oral suspension formulation of NTZ; participants 12 years and older will receive NTZ tablets.
  Nitazoxanide (NTZ): Participants 1 to 3 years old: 5 mL oral suspension (100 mg NTZ) every 12 hours for 5 days.
  Participants 4 to 11 years old: 10 mL oral suspension (200 mg NTZ) every 12 hours for 5 days.
  Participants 12 years and older: two 300-mg NTZ tablets orally twice daily for 5 days.
- Placebo: Participants will receive placebo for 5 days. Participants younger than 12 years will receive an oral suspension formulation of placebo; participants 12 years and older will receive placebo tablets.
  Placebo: Participants 1 to 3 years old: 5 mL placebo oral suspension every 12 hours for 5 days.
  Participants 4 to 11 years old: 10 mL placebo oral suspension every 12 hours for 5 days.
  Participants 12 years and older: two placebo tablets orally twice daily for 5 days.
Period: Overall Study
Arm/Group | Nitazoxanide (NTZ) | Placebo
Started | 131 | 129
Intent to Treat | 130 | 127
Completed | 117 | 121
Not Completed | 14 | 8
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 8 | 3
Not completed — Non-compliance | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis was based on the ITT population of 257 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitazoxanide (NTZ) | Placebo | Total
Number analyzed (Participants) | 130 | 127 | 257
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 67 | 64 | 131
  Between 18 and 65 years | 54 | 56 | 110
  >=65 years | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.6 (24.0) | 23.6 (24.4) | 23.1 (24.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 50 | 118
  Male | 62 | 77 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 130 | 127 | 257
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 129 | 127 | 256
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 130 | 127 | 257
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: The analysis only includes the adult (>= 18 years) population with evaluable data.
  kg/m^2
    number analyzed (Participants) | 63 | 62 | 125
    (all) | 27.2 (6.2) | 27.0 (5.6) | 27.1 (5.9)
BMI Z Score [Mean (Standard Deviation); unit: Z Score] — The Z-score indicates the number of standard deviations away from a reference population matched for age and gender. A Z-score of 0 is equal to the reference population. Negative numbers indicate BMI values lower than the reference population and positive numbers indicate values higher than the reference population. Population: The analysis only included the child (< 18 years) population with evaluable data.
  Z Score
    number analyzed (Participants) | 66 | 64 | 130
    (all) | 0.2 (2.0) | -0.6 (2.5) | -0.2 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Time to Hospital Discharge
Description: The time to hospital discharge measured through Day 28.
Time Frame: Measured through Day 28
Measure: Mean (Standard Error); unit: Days
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
Days | 7.1 (0.37) | 7.5 (0.41)
Statistical Analysis 1: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Equivalence — The equivalence margin is 1.25 Days; p = 0.5634, Fay - Shaw

2. Secondary Outcome: Number of Participants Hospitalized on Days 3, 7, 14, and 28
Description: The number of study participants (e.g., adults and children) who were hospitalized on Days 3, 7, 14, and 28.
Time Frame: Measured at Day 3, Day 7, Day 14, and Day 28
Population: Number of study participants - adults (>= 18 years) and children (< 18 years) in the Intent-to-Treat population (ITT) hospitalized by time point
Measure: Number; unit: participants
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
participants
  Day 3 | 95 | 96
  Day 7 | 39 | 38
  Day 14 | 7 | 6
  Day 28 | 3 | 2
Statistical Analysis 1: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.645, Fay - Shaw — The p-value for each time point was calculated; Day 3
Statistical Analysis 2: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.989, Fay-Shaw — The p-value for each value was calculated (Day 7)
Statistical Analysis 3: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.809, Fay-Shaw — Day 14
Statistical Analysis 4: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.671, Fay-Shaw — Day 28

3. Secondary Outcome: Number of Participants Who Died Within the First 5 Days
Description: Total Deaths of Participants, including Deaths within First 5 Days
Time Frame: Measured within First 5 Days
Population: The Adult (>=18 Years) population includes 126 participants (63 in NTZ arm; 63 in Placebo arm). The Children (<18 Years) population includes 131 participants (67 in NTZ arm; 64 in Placebo arm)
Measure: Number; unit: participants
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
participants
  Total Deaths | 2 | 1
  Deaths within the First 5 Days (Adults >=18) Years: number analyzed (Participants) | 63 | 63
  Deaths within the First 5 Days (Adults >=18) Years | 0 | 0
  Deaths within the First 5 Days (Children<18) Years: number analyzed (Participants) | 67 | 64
  Deaths within the First 5 Days (Children<18) Years | 0 | 0

4. Secondary Outcome: Number of Participants Who Experienced Clinical Symptoms
Description: Measured daily through Study Day 14 and then again on Study Day 28
Time Frame: Measured through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
Participants
  Cough | 71 | 75
  Sore Throat | 29 | 23
  Fatigue | 60 | 54
  Nasal Discharge | 40 | 25
  Difficulty Breathing | 54 | 51
  Headache | 21 | 13
  Muscle Pain | 28 | 18
  Nausea | 4 | 8
  Vomiting | 5 | 7
  Diarrhea | 4 | 5
Statistical Analysis 1: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.4277, Fay - Shaw — Cough
Statistical Analysis 2: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.4022, Fay-Shaw — Sore Throat
Statistical Analysis 3: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.5957, Fay-Shaw — Fatigue
Statistical Analysis 4: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.0446, Fay-Shaw — Nasal Discharge
Statistical Analysis 5: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.8628, Fay-Shaw — Difficulty Breathing
Statistical Analysis 6: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.16, Fay-Shaw — Headache
Statistical Analysis 7: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.1234, Fay-Shaw — Muscle Pain
Statistical Analysis 8: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.2155, Fay-Shaw — Nausea
Statistical Analysis 9: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.5176, Fay-Shaw — Vomiting
Statistical Analysis 10: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.6986, Fay-Shaw — Diarrhea

5. Secondary Outcome: Duration of Fever in Study Participants
Description: Study participants' duration (hours) of fever measured daily through Day 14 and then again on Day 28. The total duration in hours from the visit when fever was registered for the study participant until the next visit when no fever was registered for the study participant.
Time Frame: Measured each day through Day 14 and on Day 28
Measure: Mean (Standard Error); unit: hours
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
hours | 11.3 (3.55) | 20.6 (5.44)
Statistical Analysis 1: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.9850, Fay - Shaw

6. Secondary Outcome: Number of Participants Who Require Oxygen Use
Description: Number of study participants who require use of supplemental oxygen at time points (e.g., Any time, Day 0, Day 3, Day 7, Day 14, and Day 28)
Time Frame: Measured through Day 28 or participants' last day of hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
Participants
  Any Time | 119 | 118
  Day 0 | 114 | 116
  Day 3 | 74 | 80
  Day 7 | 28 | 27
  Day 14 | 6 | 5
  Day 28 | 6 | 4
Statistical Analysis 1: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.681, Fay - Shaw — Any Time
Statistical Analysis 2: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.341, Fay-Shaw — Day 0
Statistical Analysis 3: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.321, Fay-Shaw — Day 3
Statistical Analysis 4: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.957, Fay-Shaw — Day 7
Statistical Analysis 5: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.788, Fay-Shaw — Day 14
Statistical Analysis 6: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.544, Fay-Shaw — Day 28

7. Secondary Outcome: Number of Study Participants (e.g., Adult and Children) Admitted to the Intensive Care Unit (ICU) by Time Point (Anytime, Day 0, Day 3, Day 7, Day 14, Day 28)
Description: Number of study participants (e.g., adult and children) admitted to the intensive care unit (ICU) by time point (Anytime, Day 0, Day 3, Day 7, Day 14, Day 28); worst case imputed.
Time Frame: Measured through Day 28 or participants' last day in the ICU
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
Participants
  Any Time | 3 | 2
  Day 0 | 3 | 1
  Day 3 | 1 | 1
  Day 7 | 1 | 1
  Day 14 | 0 | 1
  Day 28 | 0 | 0
Statistical Analysis 1: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.671, Fay - Shaw — Any Time
Statistical Analysis 2: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.325, Fay-Shaw — Day 0
Statistical Analysis 3: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.987, Fay-Shaw — Day 3
Statistical Analysis 4: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.987, Fay-Shaw — Day 7
Statistical Analysis 5: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.311, Fay-Shaw — Day 14

8. Secondary Outcome: Study Participants (e.g., Adults, Children) Requiring Mechanical Ventilation at Study Time Points (Any Time, Day 0, Day 3, Day 7, Day 14, Day 28)
Description: Study participants (e.g., adults, children) requiring mechanical ventilation (e.g., intubation/extubation) at study time points (Any Time, Day 0, Day 3, Day 7, Day 14, Day 28); worst case imputed.
Time Frame: Measured through Day 28 or participants' last day of hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
Participants
  Any Time | 4 | 4
  Day 0 | 2 | 1
  Day 3 | 1 | 2
  Day 7 | 1 | 1
  Day 14 | 1 | 1
  Day 28 | 1 | 1
Statistical Analysis 1: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.973, Fay - Shaw — Any Time
Statistical Analysis 2: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.575, Fay-Shaw — Day 0
Statistical Analysis 3: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.548, Fay-Shaw — Day 3
Statistical Analysis 4: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.987, Fay-Shaw — Day 7
Statistical Analysis 5: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.987, Fay-Shaw — Day 14
Statistical Analysis 6: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.987, Fay-Shaw — Day 28

9. Secondary Outcome: Number of Study Participants With the Presence of Complications (Pneumonia, Respiratory Failure Requiring Mechanical Ventilation, Acute Respiratory Distress Syndrome [ARDS], Sepsis, or Bronchiolitis) During Study
Description: Number of study participants (e.g., adults and children) with the presence of a complication (pneumonia, respiratory failure requiring mechanical ventilation, acute respiratory distress syndrome [ARDS], sepsis, or bronchiolitis) during the study .
Time Frame: Measured through Day 28 or participants' last day of hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
Participants
  Pneumonia | 74 | 73
  Respiratory Failure Requiring Mechanical Vent. | 0 | 0
  Acute Respiratory Distress Syndrome (ARDS) | 6 | 6
  Sepsis | 0 | 0
  Bronchitis | 2 | 7
Statistical Analysis 1: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.928, Fay - Shaw — Pneumonia
Statistical Analysis 2: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.9669, Fay-Shaw — ARDS
Statistical Analysis 3: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.0832, Fay-Shaw — Bronchitis

10. Secondary Outcome: Duration (Days) Until Affirmative Global Assessment (e.g., Answered Yes) by Study Participants (e.g., Adults, Children)
Description: Study participant (e.g., adults and children) answers (e.g., yes) to global assessment questions measured daily through Day 14 and then again on Day 28.
Time Frame: Measured daily through Day 14 and on Day 28
Measure: Mean (Standard Error); unit: days
Groups:
- Nitazoxanide (NTZ) - Adults >=18 Years; Nitazoxanide (NTZ) - Children <18 Years: Participants will receive NTZ for 5 days. Participants younger than 12 years will receive an oral suspension formulation of NTZ; participants 12 years and older will receive NTZ tablets.
  Nitazoxanide (NTZ): Participants 1 to 3 years old: 5 mL oral suspension (100 mg NTZ) every 12 hours for 5 days.
  Participants 4 to 11 years old: 10 mL oral suspension (200 mg NTZ) every 12 hours for 5 days.
  Participants 12 years and older: two 300-mg NTZ tablets orally twice daily for 5 days.
- Placebo - Adults >=18 Years; Placebo - Children <18 Years: Participants will receive placebo for 5 days. Participants younger than 12 years will receive an oral suspension formulation of placebo; participants 12 years and older will receive placebo tablets.
  Placebo: Participants 1 to 3 years old: 5 mL placebo oral suspension every 12 hours for 5 days.
  Participants 4 to 11 years old: 10 mL placebo oral suspension every 12 hours for 5 days.
  Participants 12 years and older: two placebo tablets orally twice daily for 5 days.
Arm/Group | Nitazoxanide (NTZ) - Adults >=18 Years | Placebo - Adults >=18 Years | Nitazoxanide (NTZ) - Children <18 Years | Placebo - Children <18 Years
Number analyzed (Participants) | 63 | 63 | 67 | 64
days
  Have you felt as good as you did before? | 10.2 (1.47) | 7.0 (1.27) | 3.3 (0.40) | 3.5 (0.63)
  Are you functioning as well as you were before? | 12.6 (1.52) | 9.4 (1.38) | 3.6 (0.43) | 3.1 (0.36)
Statistical Analysis 1: Comparison: Nitazoxanide (NTZ) - Adults >=18 Years vs Placebo - Adults >=18 Years; Test type: Superiority; p = 0.0360, Fay - Shaw — Adults (>= 18 Years ) - Global Assessment: Have you felt as good as you did before you had the respiratory illness?
Statistical Analysis 2: Comparison: Nitazoxanide (NTZ) - Adults >=18 Years vs Placebo - Adults >=18 Years; Test type: Superiority; p = 0.0380, Fay-Shaw — Adults (>= 18 Years) - Global Assessment: Are you functioning as well as you were before you had the respiratory illness?
Statistical Analysis 3: Comparison: Nitazoxanide (NTZ) - Children <18 Years vs Placebo - Children <18 Years; Test type: Superiority; p = 0.5035, Fay-Shaw — Children (< 18 Years) - Global Assessment: Have you/your child felt as good as you did before you had the respiratory illness?
Statistical Analysis 4: Comparison: Nitazoxanide (NTZ) - Children <18 Years vs Placebo - Children <18 Years; Test type: Superiority; p = 0.9231, Fay-Shaw — Children (<18 Years) - Global Assessment: Are you/your child functioning as well as you/your child were before you/your child had the respiratory illness?

11. Secondary Outcome: Number of Participants Using Antibiotics/Antivirals During Hospitalization
Description: Number of study participants taking an Antibiotic or Anti-Influenza Antiviral during first 5 days of hospitalization.
Time Frame: Measured through participants' first 5 days of hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
Participants
  Antibiotic Use During First 5 Days of Hosp | 100 | 88
  Antiviral Use During First 5 Days of Hosp | 46 | 45

12. Secondary Outcome: Number of Participants Who Are Re-hospitalized Within 28 Days
Description: Number of study participants (e.g., adults and children) who were re-hospitalized within 28 days (e.g., days from randomization).
Time Frame: Measured through Day 28
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
participants
  Adults >=18 Years: number analyzed (Participants) | 63 | 63
  Adults >=18 Years | 1 | 2
  Children >18 Years: number analyzed (Participants) | 67 | 64
  Children >18 Years | 1 | 2

13. Secondary Outcome: Use of Systemic Corticosteroids
Description: Number of study participants taking Systemic Steroids during first 5 days.
Time Frame: Measured within First 5 Days
Population: The analysis was based on the Intent to Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
Participants
  Subjects Taking Systemic Steroids - First 5 Days | 78 | 70
  DESMOPRESSIN | 0 | 1
  DEXAMETHASONE | 4 | 5
  GLUCOCORTICOIDS (Fluticasone/Vilanterol) | 0 | 1
  HYDROCORTISONE | 5 | 3
  LEVOTHYROXINE | 6 | 8
  LEVOTHYROXINE SODIUM | 1 | 1
  METHYLPREDNISOLONE | 35 | 26
  NOVOTHYRAL | 0 | 1
  PREDNISONE | 43 | 35

14. Secondary Outcome: Presence of Virus on Nasopharyngeal (NP) Swab at Day 3 (Same Virus as Day 0)
Description: Study participants with Detectable Virus on nasopharyngeal (NP) swab at Baseline and at Day 3.
Time Frame: Measured through Day 3
Population: Efficacy analysis of Intent to Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 79 | 89
Participants
  No Detectable Virus on Day 3 | 17 | 19
  Same Detectable Virus on Day 3 | 56 | 61
  Different Detectable Virus on Day 3 | 6 | 9
Statistical Analysis 1: Comparison: Nitazoxanide (NTZ) vs Placebo; Test type: Superiority; p = 0.9785, Fay-Shaw — No Detectable Virus on Day 3

15. Secondary Outcome: Number of Participants Reporting Adverse Events (AEs)
Description: Number of study participants with at least one Adverse Event During Study Duration
Time Frame: Measured through Day 28 or participants' last day of hospitalization
Population: Analysis was based on the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
Participants | 83 | 80

16. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: Number of study participants (e.g., adults and children) reporting at least one serious adverse events (SAEs).
Time Frame: Measured through Day 28 or participants' last day of hospitalization
Population: The analysis is based on the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
Participants | 6 | 3

17. Secondary Outcome: Chemistry Laboratory Assessments (Creatinine, Total Bilirubin) on Days 3, 7, and 28
Description: Laboratory values for chemistry laboratory assessments (e.g., Creatinine and Total Bilirubin) on Days 3, 7, and 28.
Time Frame: Measured on Day 3, Day, 7 and Day 28
Population: This analysis was based on the Intent to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
mg/dL
  Creatinine (mg/dL): Day 3 | 0.5 (0.3) | 0.6 (0.4)
  Creatinine (mg/dL): Day 7 | 1.1 (5.3) | 0.6 (0.3)
  Creatinine (mg/dL): Day 28 | 0.6 (1.1) | 0.6 (0.4)
  Total Bilirubin (mg/dL): Day 3 | 0.6 (0.4) | 0.5 (0.3)
  Total Bilirubin (mg/dL): Day 7 | 1.0 (4.6) | 0.5 (0.3)
  Total Bilirubin (mg/dL): Day 28 | 0.6 (0.3) | 0.6 (0.3)

18. Secondary Outcome: Chemistry Laboratory Assessments (ALT, AST, LDH) on Days 3, 7, and 28
Description: Chemistry laboratory assessments (e.g., ALT, AST, and LDH) on Days 3, 7, and 28.
Time Frame: Measured on Day 3, Day 7, and Day 28
Population: This analysis was based on the Intent to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
U/L
  ALT (SGPT) (U/L): Day 3 | 32.7 (24.6) | 30.9 (27.2)
  ALT (SGPT) (U/L): Day 7 | 33.1 (20.5) | 35.1 (28.7)
  ALT (SGPT) (U/L): Day 28 | 26.7 (15.4) | 27.4 (16.8)
  AST (SGOT) (U/L): Day 3 | 32.7 (19.4) | 36.1 (30.4)
  AST (SGOT) (U/L): Day 7 | 33.2 (20.2) | 33.2 (19.0)
  AST (SGOT) (U/L): Day 28 | 33.0 (20.0) | 31.8 (18.5)
  LDH (U/L): Day 3 | 248.1 (164.8) | 266.8 (180.0)
  LDH (U/L): Day 7 | 250.3 (151.4) | 255.2 (150.8)
  LDH (U/L): Day 28 | 241.8 (141.6) | 249.7 (151.3)

19. Secondary Outcome: Chemistry Laboratory Assessment (CRP) on Days 3, 7, and 28
Description: Lab Values for chemistry laboratory assessment (e.g., CRP) on Days 3, 7, and 28.
Time Frame: Measured on Day 3, Day, 7 and Day 28
Population: This analysis was based on the Intent to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
mg/L
  CRP (mg/L): Day 3 | 2.3 (4.1) | 2.2 (3.4)
  CRP (mg/L): Day 7 | 1.2 (3.3) | 1.1 (2.4)
  CRP (mg/L): Day 28 | 1.1 (3.7) | 0.5 (0.7)

20. Secondary Outcome: Hematologic Laboratory Assessments (Neutrophils, Lymphocytes, Eosinophils, and Hematocrit) on Days 3, 7, and 28
Description: Hematology laboratory assessments (e.g., Neutrophils, Lymphocytes, Eosinophils, and Hematocrit) on Days 3, 7, and 28.
Time Frame: Measured on Day 3, Day, 7 and Day 28
Population: This analysis was based on the Intent to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: percentage of blood
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
percentage of blood
  Neutrophils (%): Day 3 | 59.1 (19.8) | 55.9 (19.3)
  Neutrophils (%): Day 7 | 52.4 (21.0) | 52.3 (17.0)
  Neutrophils (%): Day 28 | 51.4 (16.6) | 49.8 (17.2)
  Lymphocytes (%): Day 3 | 31.6 (17.5) | 33.4 (17.0)
  Lymphocytes (%): Day 7 | 36.5 (19.3) | 36.7 (16.0)
  Lymphocytes (%): Day 28 | 36.1 (15.2) | 37.5 (16.9)
  Eosinophils (%): Day 3 | 1.5 (2.2) | 2.3 (5.2)
  Eosinophils (%): Day 7 | 2.3 (1.9) | 2.6 (2.7)
  Eosinophils (%): Day 28 | 3.8 (4.3) | 3.6 (4.1)
  Hematocrit (%): Day 3 | 41.3 (5.6) | 40.6 (6.1)
  Hematocrit (%): Day 7 | 40.7 (5.3) | 40.9 (6.1)
  Hematocrit (%): Day 28 | 41.2 (4.6) | 41.7 (6.1)

21. Secondary Outcome: Hematologic Laboratory Assessment (Hemoglobin) on Days 3, 7, and 28
Description: Hematology laboratory assessment (e.g., Hemoglobin) on Days 3, 7, and 28.
Time Frame: Measured on Day 3, Day, 7 and Day 28
Population: This analysis was based on the Intent to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
g/dL
  Hemoglobin (g/dL): Day 3 | 13.5 (1.8) | 13.2 (2.0)
  Hemoglobin (g/dL): Day 7 | 13.5 (1.7) | 13.4 (2.1)
  Hemoglobin (g/dL): Day 28 | 13.6 (1.5) | 13.6 (2.0)

22. Secondary Outcome: Hematologic Laboratory Assessments (WBC, Platelets) on Days 3, 7, and 28
Description: Lab values for hematology laboratory assessments (e.g., WBC and Platelets) on Days 3, 7, and 28.
Time Frame: Measured on Day 3, Day, 7 and Day 28
Population: This analysis was based on the Intent to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: 10^3 cells/mcL
Arm/Group | Nitazoxanide (NTZ) | Placebo
Number analyzed (Participants) | 130 | 127
10^3 cells/mcL
  WBC (10^3 cells/mcL): Day 3 | 9.0 (3.9) | 8.2 (3.4)
  WBC (10^3 cells/mcL): Day 7 | 9.8 (3.9) | 9.1 (3.8)
  WBC (10^3 cells/mcL): Day 28 | 8.1 (3.1) | 8.2 (3.3)
  Platelets (10^3 cells/mcL): Day 3 | 301.3 (123.5) | 295.8 (113.7)
  Platelets (10^3 cells/mcL): Day 7 | 364.7 (155.9) | 393.3 (191.2)
  Platelets (10^3 cells/mcL): Day 28 | 269.0 (85.5) | 267.5 (110.9)

ADVERSE EVENTS:
Time Frame: AEs were recorded for each subject starting at completing the Informed Consent process and continuing until the subject completed study, or until resolution of the adverse event as recorded by the clinical site (up to Day 28).
Description: The definition of AEs and SAEs used to collect AE event information for this study does not differ from the clinicaltrials.gov definitions. The study Investigators evaluated AEs with respect to Seriousness (as per the protocol), Severity (grading), and Causality according to the "DAIDS (Division of AIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events" Version 1.0, December 2004: (Clarification August 2009)
Arm/Group | Nitazoxanide (NTZ) | Placebo
All-Cause Mortality (participants affected / at risk) | 2/130 | 1/127
Serious Adverse Events (participants affected / at risk) | 6/130 | 3/127
Other Adverse Events (participants affected / at risk) | 26/130 | 26/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitazoxanide (NTZ) (N=130) | Placebo (N=127)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia Viral (Infections and infestations) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 1 (1) | 1 (1)
Immune Reconstitution Inflammatory Syndrome Associated Kaposi's Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitazoxanide (NTZ) (N=130) | Placebo (N=127)
Vomitting (Gastrointestinal disorders) | 8 (9) | 14 (14) — MedDRA System Organ Class and Preferred term.
Pyrexia (General disorders) | 8 (8) | 5 (5) — MedDRA System Organ Class and Preferred Term.
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 7 (7) — MedDRA System Organ Class and Preferred Term.

LIMITATIONS AND CAVEATS:
There were no significant limitations of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT02057757/SAP_000.pdf
  • Study Protocol (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT02057757/Prot_001.pdf